CLINICAL TRIAL: NCT02088970
Title: Safety and Efficacity of Corneal Collagen Crosslinking in Infectious Keratitis (Bacterial and Fungal ): Randomized,Controlled, Prospective Study.
Brief Title: Safety and Efficacity of Corneal Collagen Crosslinking in Infectious Keratitis (Bacterial and Fungal ): Randomized,Controlled, Prospective Study. (CXL)
Acronym: CXL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties in reaching the desired number of patients and intermediate analysis leading to discontinuation of the study.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC14_0004
Record Dates: First submitted 2014-03-13; First posted 2014-03-17 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Bacterial Keratitis; Fungal Keratitis
Keywords: Infectious keratitis; Corneal cross linking; Topical antibiotics
MeSH Terms: interventions — Chromatin Immunoprecipitation Sequencing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- antibiotic treatment alone (Active Comparator)
  Interventions: Drug: antibiotic treatment
- Crosslinking + Antibiotic (Experimental): The procedure of the cross linking is standard:combined riboflavin(Ricrolin®)-ultraviolet type A rays (UVA) collagen cross-linking. Radiant energy was 3 milliwatts/cm2 or 5.4 joule/cm2 for a 30-minute exposure irradiation of the cornea.
  Patients are checked every days during the hospitalisation and one week, one month and 3 months after the hospitalisation.
  Interventions: Device: Crosslinking; Drug: antibiotic treatment

INTERVENTIONS:
Device: Crosslinking — The procedure of the cross linking is standard:combined riboflavin(Ricrolin®)-ultraviolet type A rays (UVA) collagen cross-linking. Radiant energy was 3 milliwatts/cm2 or 5.4 joule/cm2 for a 30-minute exposure irradiation of the cornea.
  Patients are checked every days during the hospitalisation and one week, one month and 3 months after the hospitalisation.
  Other Names: Riboflavine 0,1%.; Ricrolin.; CE 0037.; médical device class IIb.; Manufacter : SOOFT Distributor : Horus pharma.; transmitter UV-A :; Model : Vega, CBM X Linker. (CSO, Florence, Italie)
  Arms: Crosslinking + Antibiotic
Drug: antibiotic treatment — If not the contact lens wearer -> Cocci Gram positive cocci
  * Vancomycin + Fortum
  If contact lens wearer -> Gram negative bacillus
  * Fortum + Amiklin
  If corticosteroids, immunosuppression, latent evolution -> Fungus.
  = Fortum + vancomycin + Fungizone

SUMMARY:
The corneal collagen cross linking is currently used in the treatment of keratoconus but this procedure has also a sterilizing non-specific effect on bacteria and fungus. So the corneal cross linking in association with the antibiotic treatment could result in a reduction of the duration of epithelial complete healing of the cornea.

ELIGIBILITY:
Inclusion Criteria:

* Infectious bacterial or fungal keratitis with : size > 2mm or within the central corneal area ( 3mm of the visual axis ) or with a reaction in anterior chamber.
* Being major responsible.
* Agreement in writing to participate in the study.
* Being affiliated to a national insurance scheme.

Exclusion Criteria:

* Present an infectious keratitis without all the previous criteria.
* Herpes or acanthamoeba keratitis
* preperforated or perforated cornea.

General criteria:

* Pregnant woman.
* Minors(miners).
* Adults under guardianship.
* Patient can not be followed during 3 necessary months.
* French speaking patient.
* Unaffiliated patient in a national insurance scheme.
* HIV infected patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Duration of corneal complete epithelial healing in days. | 3 months

SECONDARY OUTCOMES:
Size of the corneal scar | 3months
  Size of the corneal scar at 3months expressed in % of the initial size of the corneal ulcer.
Corneal thinning | 3 months
  Corneal thinning estimated by Anterior segment optical coherence tomography at 3 months, expressed in microns.
Gain of visual acuity | 3 months
  Gain of visual acuity, corresponding to the difference between the initial visual acuity and the 3months one. The visual acuity is measured with monoyer scale and converted in log Mar.

CONTACTS AND LOCATIONS:
Locations (1):
- Orignac, Nantes, France

REFERENCES:
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558